CLINICAL TRIAL: NCT06721585
Title: A Randomized, Placebo-controlled, Double-blinded Trial of the Safety and Efficacy of Tecovirimat for the Treatment of Adult and Pediatric Patients With Monkeypox Virus Disease - Extension Amendment
Brief Title: Tecovirimat for Treatment of Monkeypox Virus - Study Extension Providing Standard of Care Only
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Other Study IDs: PALM007-Ext
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Mpox (Monkeypox)
Keywords: Mpox; MPXV; Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, mouth swabs, skin lesion swabs, , skin biopsies, conjunctival swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Open-access tecovirimat plus SOC for mpox: Participants are provided SOC as well as open-access tecovirimat. Tecovirimat capsules are administered orally to participants for 14 days based on participant weight.
  Closed to new participants in August 2024.
  Interventions: Drug: Tecovirimat Oral Capsule [Tpoxx]; Other: Standard of Care (SOC)
- Standard of care for mpox: Participants are provided SOC for mpox.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Tecovirimat Oral Capsule [Tpoxx] — Tecovirimat Oral Capsule 200 mg capsules
  Number of capsules and frequency of dosage will be based on participant weight:
  * ≥120 kg: three capsules three times a day (total daily tecovirimat dose: 1,800 mg)
  * 40 to <120 kg: three capsules twice a day (total daily tecovirimat dose: 1,200 mg)
  * 25 to <40 kg: two capsules twice a day (total daily tecovirimat dose: 800 mg)
  * 13 to <25 kg: one capsule twice a day (total daily tecovirimat dose: 400 mg)
  * 6 to <13 kg: ½ the contents of a capsule twice daily (total daily tecovirimat dose: 200 mg)
  * 3 to <6 kg: ¼ the contents of a capsule twice daily (total daily tecovirimat dose: 100 mg)
  Other Names: TPOXX
  Groups: Open-access tecovirimat plus SOC for mpox
Other: Standard of Care (SOC) — Participants are provided SOC for mpox

SUMMARY:
The purpose of the PALM007 extension is to further characterize the clinical and natural history of mpox, and to provide standard of care (SOC) during the ongoing outbreaks.

DETAILED DESCRIPTION:
This open-label extension to the PALM007 protocol began in July 2024 after enrollment into the main study ended. It will further clinically characterize the natural history of mpox, and continue to identify recrudescent cases. Participants were initially provided SOC as well as open-access tecovirimat. The results of PALM007 were unblinded in August 2024, and although no safety concerns were observed with tecovirimat use, efficacy, defined by improvement in days to complete mpox skin lesion resolution, was not observed for tecovirimat compared to placebo. Therefore, the administration of tecovirimat in the extension amendment was discontinued in early August 2024, once these results were known, and only SOC continues to be provided.

Participants are admitted to the hospital and receive SOC for mpox until they have recovered. Recovery is defined as resolution of all lesions and a negative blood test for MPXV. Participants will remain on study through day 59 but will not have a scheduled study visit unless they present with new mpox symptoms. Sick visits will be available for participants who reach full body lesion resolution but subsequently develop at least 1 new lesion consistent with mpox after discharge and on or before day 59, at which time viral PCR and clinical laboratory testing will be performed and participants will be offered standard of care.

Initially, all participants presenting with mpox were eligible to enroll in this extension, regardless of disease severity. As of 05May2025, only patients with severe disease, defined as the presence of any of the following: flat lesions, pregnancy (due to risk for serious complications), suspected sickle cell disease, or severe clinical disease will be enrolled.

ELIGIBILITY:
This study has no age restriction

Inclusion Criteria:

1. Laboratory-confirmed mpox infection as determined by PCR obtained from blood, oropharynx, or skin lesion within 48 hours of screening
2. Mpox illness of any duration provided that the patient has at least one active, not yet scabbed, lesion
3. Stated willingness to comply with all study procedures (including required inpatient stay) and availability for the duration of the study
4. Ability to provide informed consent personally or by a legally or culturally acceptable representative if the patient is unable to do so
5. Severe disease, defined as the presence of at least one of the following:

   1. Flat lesions (flat and soft lesions; no pustules or vesicles visible to the eye)
   2. Pregnancy (due to risk of serious complication)
   3. Suspected sickle cell disease
   4. Severe clinical disease, defined as having at least 3 of the following:

      * Lesion count greater than 250
      * Fever for greater than 48 hours
      * Hypotension (systolic blood pressure less than 90 mmHg or diastolic blood pressure less than 60 mmHg)
      * Pallor
      * Respiratory distress
      * Altered mental status
      * Extreme lethargy
      * Painful oral lesions making oral intake difficult
      * Difficulty peeing or pooping due to painful lesions
      * Painful lesions on hands and feet
      * Tachycardia (heart rate greater than 100 beats per minute)
      * Diarrhea (greater than or equal to 3 liquid stools per 24 hours)

Exclusion Criteria:

1. Severe anemia, defined as hemoglobin less than 7 g/dL
2. Current or planned use of another investigational drug at any point during study participation
3. Patients who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with laboratory-confirmed monkeypox virus (MPXV) disease at participating sites in the Democratic Republic of Congo
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Time to lesion resolution | up to day 28
  Number of days to the first day on which all lesions on the total body are scabbed or desquamated or a new layer of epidermis has formed.

SECONDARY OUTCOMES:
Time to lesion resolution for participants with symptom onset less than or equal to 7 days enrollment | up to day 28
  Number of days to the first day on which all lesions on the total body are scabbed or desquamated or a new layer of epidermis has formed.
Time to lesion resolution for participants with symptom onset greater than 7 days before enrollment | up to day 28
  Number of days to the first day on which all lesions on the total body are scabbed or desquamated or a new layer of epidermis has formed.
Number of participants that develop at least 1 new mpox lesion after discharge | up to day 59
  Number of participants who reach full body lesion resolution, and develop at least 1 new lesion after discharge
Mortality within the first 28 days post-enrollment | up to day 28
  Number of deaths post-enrollment
Number of days to participant death | up to day 59
  Number of days post-enrollment
Frequency of solicited clinical symptoms | up to day 59
  Clinical symptoms defined as: nausea, vomiting, abdominal pain, diarrhea, anorexia, cough, lymphadenopathy, dysphagia, sore throat, muscle aches, fatigue/lack of energy, fever, chills, night sweats, headache, ocular lesions, eye pain, change in vision, buccal ulcers, nasal congestion, cough, joint pain, pain with urination, painful skin lesions, pruritic skin lesions.
Duration of solicited clinical symptoms | up to day 59
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Muyembe-Tamfum, MD PhD, Principal Investigator — Kinshasa University
Locations (2):
- Democratic Republic of the Congo (2):
  - L'Hôpital Général de Référence de Kole, Kole
  - L'Hôpital Général de Référence de Tunda, Tunda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PALM 007 Record NCT05559099 — https://clinicaltrials.gov/study/NCT05559099

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT06721585/ICF_000.pdf